CLINICAL TRIAL: NCT05909774
Title: Assessment of the Interest of the Atalante Device for Patients With Manual Wheelchairs
Acronym: M1-M2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-A01257-44
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Complete Motor Paraplegia
Keywords: exoskeleton; paraplegia; rehabilitation
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, comparative, randomized cross-over study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exoskeleton second (Experimental): This group first perform tests without Atalante exoskeleton and secondly with Atalante exoskeleton. A second randomization is performed inside each group, with half of the patients first performing walk test with the "Continuous" walk and then with the "Push & Swing" walk, and the other half doing the opposite.
  Interventions: Device: Test with Atalante exoskeleton in "continuous walk" type
- Exoskeleton first (Active Comparator): This group first perform tests with Atalante exoskeleton and secondly without Atalante exoskeleton. A second randomization is performed inside each group, with half of the patients first performing walk test with the "Continuous" walk and then with the "Push & Swing" walk, and the other half doing the opposite.
  Interventions: Device: Test with Atalante exoskeleton in "continuous walk" type

INTERVENTIONS:
Device: Test with Atalante exoskeleton in "continuous walk" type — The "continuous" walk is smoother and more physiologic than the "push and swing" walk
  Other Names: Test with Atalante exoskeleton in "push and swing" walk type

SUMMARY:
The loss of standing and walking capabilities in a paraplegic person is most often the result of damage to the spinal cord, either traumatic (accidental) or pathological and has both a somatic and a psychological impact on the quality of life, the risk of depression, and the difficulty of socio-professional reintegration in a society that is not adapted to people with disabilities.

A motorized mechanical exoskeleton is an external device intended to compensate for a muscular or neurological deficiency enabling paraplegics to stand and walk again. The Atalante exoskeleton, designed by Wandercraft company allows patients to stand upright and walk without the aid of crutches.

This early study was the first clinical investigation of the Atalante exoskeleton performed early in the development. It was used to evaluate the device design concept with respect to initial clinical safety and device functionality and guided further device modifications.

DETAILED DESCRIPTION:
The aim of this study was to test the use of the Atalante exoskeleton on 10 patients with complete motor paraplegia (ASIA A and B) with a level of injury between T6 and S1.

In this multi-centric clinical trial, patients were asked to perform between 1 and 2 days of training with Atalante exoskeleton including device training and evaluations (up to 9 hours of training and 3 hours of evaluation per patient).

The primary objective of this study was to assess patients' ability to walk straight- for 10 meters with the Atalante exoskeleton during 10-meters walk test (10MWT).

Within-group differences between the Atalante exoskeleton and the usual walking aid used by the patient in the success rate of the 10MWT were compared by a McNemar test.

The secondary objectives focused on performance evaluation with the Atalante exoskeleton. The assessments performed were:

1. Assessment of the superiority of the Atalante exoskeleton compared to the usual aid walking assistance used by the patient on the walking, verticalization (or sit-to-stand), static and dynamic balance ability
2. Assessment of the static and dynamic postural stability of the subject with the Atalante exoskeleton by observation of center of pressure displacement and velocity
3. Assessment of the perceived effort by the patient
4. Assessment of perceived safety by the patient
5. Assessment of the overall satisfaction of patients after using the exoskeleton
6. Comparison of the two types of walk on walking ability, perceived effort, and safety

ELIGIBILITY:
Inclusion Criteria:

* Under 60 years of age
* Daily and autonomous use of wheelchair
* Paraplegia with level of injury between T6 and S1
* Patient unable to walk, neither during physiotherapy session nor in a daily routine
* Patient with cognitive capacities: able to understand oral and/or written instructions, as well as instructions given by demonstration
* Able to use their upper limbs
* Can be verticalized
* Patient with a health care insurance
* Patient having given his/her written consent
* Joints amplitudes compatible with the use of the exoskeleton:
* Hip: Flexion>115°; Extension>15°; Abduction>17°; Adduction >10°; Medial rotation>35°; Internal rotation>10°
* Knee: Flexion>105°; Extension> -5°
* Ankle: Flexion>0°; Extension>9°; Supination>18°; Pronation>18°

Exclusion Criteria:

* Severe or complete deficiency of the upper limbs
* Bad control of the trunk
* Vestibular disorder (loss of balance, dizziness, …) when placed in the vertical position
* Upper limbs involuntary shivers and/or movements
* Pregnant women
* A lower or upper limb amputated
* Epilepsy
* Patient carrying an active implantable medical device

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to assess patients' ability to walk straight- for 10 meters with the Atalante exoskeleton during 10-meters walk test (10MWT). | Day 2
  Within-group differences between the Atalante exoskeleton and the usual walking aid used by the patient in the success rate of the 10MWT were compared by a McNemar test.

SECONDARY OUTCOMES:
Assessment of the superiority of the Atalante exoskeleton compared to the usual aid | Day 2
  Evaluation of walking ability through a 10mWT
Assessment of the superiority of the Atalante exoskeleton compared to the usual aid | Day 2
  Evaluation of verticalization ability through a success/failure test in a verticalization test (sit-to-stand movement)
Assessment of the superiority of the Atalante exoskeleton compared to the usual aid | Day 2
  Evaluation of static balance through a success failure in a static standing test without support from the operator (3 x 30s in a static standing position)
Assessment of the superiority of the Atalante exoskeleton compared to the usual aid | Day 2
  Evaluation of dynamic balance through a success/failure in a pointing test performed in a standing position without support from the operator (3 pointing sequences)
Assessment of the static and dynamic postural stability | Day 2
  Static balance test with measurement of center of pressure displacement
Assessment of the static and dynamic postural stability | Day 2
  Dynamic balance test with measurement of the average surface area under the (Center of Pressure position, Center of Pressure velocity) curve
Assessment of the perceived effort by the patient | Day 2
  Evaluation of perceived effort by the patient through a Borg CR-10 scale
Assessment of perceived safety by the patient | Day 2
  Evaluation of perceived safety by the patient through a 7-point Likert scale
Assessment of the overall satisfaction of patients after using the exoskeleton | Day 2
  Assessment of the patient overall satisfaction through a 7-point Likert scale
Comparison of the two types of walk | Day 2
  Comparison of the two types of walk on walking ability through the 10mWT
Comparison of the two types of walk | Day 2
  Comparison of the two types of walk on perceived effort during the 10mWT through a Borg CR-10 Scale
Comparison of the two types of walk | Day 2
  Comparison of the two types of walk on perceived safety during the 10mWT through a 7-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Albert, MD, Principal Investigator — COS CMPR de Bobigny
Locations (1):
- CEREMH (Centre de ressources et d'innovation mobilité handicap), Vélizy-Villacoublay, France

IPD SHARING:
Plan to Share IPD: No